CLINICAL TRIAL: NCT00177138
Title: Use of Campath for Induction and Maintenance Therapy in Pancreas After Kidney Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The clinical use of Campath for transplant patients was temporarily suspended.
Sponsor: University of Minnesota (Other)
Collaborators: Bayer (Industry); Gruessner, Rainer, MD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0308M51264; Berlex Study No. 107.G0001
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Campath Study; Pancreas After Kidney Transplantation; Alemtuzumab
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tacrolimus; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 2 (Active Comparator): Tacrolimus/MMF/TMG
  Interventions: Drug: Tacrolimus
- Group 1 (Experimental): Campath/MMF/TMG
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Tacrolimus — Starting POD #1 0.06 mg/kg/day in 2 divided doses;
  Arms: Group 2
Drug: Alemtuzumab — 30 mg IV intra-op and POD #12; then 30 mg IV >monthly for 1 year (only if ALC>200 mm, up to a total of 10 doses in year)
  Arms: Group 1

SUMMARY:
This is a single center, prospective, open-label, randomized trial at the University of Minnesota Medical Center,Fairview.

Primary objectives are to determine if rejection episodes and loss rates, graft survival, level of renal graft function, and patient survival rates with a Campath/MMF-based (Group 1) immunosuppressive protocol are lower than, or equal to, our protocol using thymoglobulin, tacrolimus, and MMF (Group 2).

This study will investigate the first protocol that is both steroid-free and calcineurin inhibitor-free in pancreas after kidney transplant recipients.

DETAILED DESCRIPTION:
Secondary objectives of the study are:

1. Compare the side effects of the immunosuppressive medications between both groups. This will include anaphylactic reactions, GI side-effects, bone marrow suppression, renal dysfunction, hypertension, hyperglycemic effects, and effects on lipid profile.
2. Compare the incidence of infections between both groups.

Comparison parameters are:

1. Pancreas and kidney graft failure
2. Patient death
3. Clinical and biopsy documented rejection episodes
4. Patient dropout (non-compliance with the study protocol)
5. Kidney function as assessed by creatinine clearance or biopsy
6. Need to change immunosuppression regimen
7. Quality-adjusted Life Years

ELIGIBILITY:
Inclusion Criteria:

1. Previous kidney transplant from a living or deceased donor and a deceased- donor pancreas transplant.
2. Recipient age 18-60 years
3. Donor age 10-59 years
4. Females of childbearing potential should have a negative pregnancy test, and agree to practice birth control for the duration of the study.
5. Enteric or bladder drained pancreas transplant.

   -

Exclusion Criteria:

1. Use of an investigational drug in the last 1-year.
2. Positive T or B cell crossmatch.
3. WBC<3000 at enrollment
4. Platelet count <50,000 at enrollment
5. History of malignancy (exclusive of minor skin cancers)
6. Inability to give informed consent
7. Systemic infections
8. Major active or chronic infections, including documented HIV infection (by any licensed ELISA and confirmation by Western Blot).
9. Serology negative for EBV pre-transplant.
10. No other previous organ transplants other than pancreas and/or kidney. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2004-07; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Time-to-event analysis will be used to analyze categorical end points that include graft failure, patient survival, biopsy documented rejection episode and non-compliance. | 2 years

SECONDARY OUTCOMES:
The continuous outcome variable, weekly or bi-weekly serum creatinine levels, will be analyzed using a two-way repeated-measures analysis of variance. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rainer W Gruessner, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota-Fairview, Minneapolis, Minnesota, United States